CLINICAL TRIAL: NCT04867265
Title: Mouth-to-mouth Ventilation Efficiency Through Breathable Self-sterilizing Respirator During BLS in COVID-19 Pandemic: a Crossover Simulation-based Study
Brief Title: Mouth-to-mouth Ventilation Efficiency Through Breathable Self-sterilizing Respirator During BLS in COVID-19 Pandemic
Acronym: MOVERESP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brno University Hospital (Other)
Collaborators: Masaryk University (Other)
Responsible Party: Principal Investigator, Petr Štourač, MD, Clinical Professor, Brno University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: SIMU 1 2021
Record Dates: First submitted 2021-04-26; First posted 2021-04-30 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-06

CONDITIONS: Ventilation During Resuscitation
Keywords: Basic life support; COVID-19; Self-sterilizing nanofiber respirator; Mouth-to-mouth ventilation; Efficiency
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Medical students trained as BLS providers (first group) and Medical student trained as teachers will perform mouth-to-mouth ventilation in 3 case scenarios on 3 different mannequins.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Professional Adult Medium Skin CPR-AED Training Manikin with CPR Monitor (Prestan) (Active Comparator): medical students trained BLS trainers and medical students trained in BLS will provide 2 minutes cycle of BLS according to ERC guidelines 2021 wearing the breathable self-sterilizing nanofiber respirators with accelerated copper
  Interventions: Procedure: Mout-to-mouth ventilation
- Resusci Anne QCPR AED (Laerdal) (Active Comparator): medical students trained BLS trainers and medical students trained in BLS will provide 2 minutes cycle of BLS according to ERC guidelines 2021 wearing the breathable self-sterilizing nanofiber respirators with accelerated copper
  Interventions: Procedure: Mout-to-mouth ventilation; Procedure: Mout-to-mouth ventilation with quantitative analysis
- Resusci Baby QCPR (Laerdal) (Active Comparator): medical students trained BLS trainers and medical students trained in BLS will provide 2 minutes cycle of BLS according to ERC guidelines 2021 wearing the breathable self-sterilizing nanofiber respirators with accelerated copper
  Interventions: Procedure: Mout-to-mouth ventilation; Procedure: Mout-to-mouth ventilation with quantitative analysis

INTERVENTIONS:
Procedure: Mout-to-mouth ventilation — we will record the visibility of chest rising
Procedure: Mout-to-mouth ventilation with quantitative analysis — we will record the visibility of chest rising, review the ventilation metrics and evaluate each rescue breath in QCPR Skill Reporter
  Other Names: Mout-to-mouth ventilation
  Arms: Resusci Anne QCPR AED (Laerdal); Resusci Baby QCPR (Laerdal)

SUMMARY:
Complex practical BLS training have been stopped all over the world due to COVID-19 pandemic in 2020. While launching the new Simulation Centre at Medical Faculty of Masaryk University in Brno, Czech Republic, teachers and students have been dealing with the risk of COVID-19 transmission during the simulation training. One of the highest risks for the transfer of COVID-19 between the medical students is during the mouth-to-mouth ventilation training in BLS.

It has been assumed that rescuers during BLS simulation training with use of breathable nanofiber respirator with layers with accelerated copper can provide efficient mouth-to-mouth rescue breaths to the mannequin in compliance with safety rules.

DETAILED DESCRIPTION:
The main aim of this study is to assess the efficiency of mouth-to-mouth ventilation through breathable self-sterilizing nanofiber respirators with accelerated copper in COVID-19 pandemic time. 100 volunteers (medical students trained as BLS trainers an medical students trained in BLS) will provide 2 minutes cycle of BLS according to European Resuscitation Council (ERC) guidelines 2021 wearing the breathable self-sterilizing nanofiber respirators with accelerated copper in three different mannequins: Professional Adult Medium Skin CPR-AED Training Manikin with CPR Monitor (Prestan), Resusci Anne QCPR AED (Laerdal), Resusci Baby QCPR (Laerdal). The mannequin will be utilised in a randomised order. The efficiency of mouth-to-mouth rescue breaths as "visible breath " and "not visible breath" will be recorded. In first BLS mannequin, the visibility of chest rising by the observer will be recorded. In two other mannequins, the ventilation metrics and each rescue breath evaluation in QCPR Skill Reporter will be recorded. Overall, 3 levels of visible breath according to the relation to set optimal breath volume (400 to 600 mL in adult, 30 to 50 mL in infant): low volume breath (below 400ml in adults and below 30ml in infant), optimal volume breath (between 400-600ml in adult and between 30-50 ml in infant), high volume breath (over 600ml in adult and over 50ml in infant) will be evaluated. For the primary analysis of efficiency of mouth-to-mouth ventilation, data from all three mannequins using outcome No breath / Visible breath will be evaluated. Secondary analysis will utilize data from two mannequins where detailed stratification No Breath / low / optimal / high Visible breath is possible. The mean volume of rescue breaths in the 2-minute cycle, average pause, longest pause, success in achieving the optimal breath volume, adverse events will be recorded. Regarding the technique of provided mouth-to-mouth ventilation, head tilt in adult or neutral position in infant and pinching of the nose will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* medical students trained in BLS as BLS trainers
* medical students trained in BLS

Exclusion Criteria:

* refusing to participate
* non-medical students

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2021-06-02 (Actual); Study Completion 2021-06-02 (Actual)

PRIMARY OUTCOMES:
Mouth-to-mouth ventilation effectivity | During 2 minute basic life support
  data from all three mannequins using variables as: No breath (chest not rising) or Visible breath (chest rising) value will be used to evaluate the overall efficacy of mouth-to-mouth ventilation

SECONDARY OUTCOMES:
mouth-to-mouth ventilation volumetric analysis | During 2 minute basic life support
  quantitative data (inspiratory volume) from two mannequins (ResusciAnne, ReusciBaby) using no breath, low, optimal, high volume breath will be evaluated
medical students trained as BLS trainers versus medical students trained in BLS mouth-to-mouth breathing efficacy | During 2 minute basic life support
  Overall efficacy of medical students trained as BLS trainers versus medical students trained in BLS will be compared taking into account no breath (chest not rising during breathnig) vs. visible breath (chest rising) on all three mannequins will be evaluated
Overall quantitative volumetric efficacy of mouth-to-mouth breathing between the medical students trained as BLS trainers versus medical students trained in BLS | During 2 minute basic life support
  Overall quantitative efficacy of mouth-to-mouth breathing of medical students trained as BLS trainers versus medical students trained in BLS will be compared taking into account no breath vs. low vs. optimal vs. high volume breath on two mannequins with the possibility of quantitative analysis (ResusiceAnne, ResusciBaby)
Correct head position incidence | During 2 minute basic life support
  The head position of the mannequin will be recorded by the observer and compared to the recommended position for the age of the patient
The incidence of ventilation without pinched nose | During 2 minute basic life support
  The incidence of ventilation without pinched nose will be recorded by the observer
Mean breath volume | During 2 minute basic life support
  Mean breath volume during mouth-to-mouth ventilation will be recorded
No-flow interval characteristics | During 2 minute basic life support
  Mean pause and the longest pause in the 2 minutes cycle of basic life support
Adverse events incidence | During 2 minute basic life support
  Incidence of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Martina Kosinova, assoc. prof. MD., Ph.D., Principal Investigator — Faculty of medicince Masaryk University and University Hospital Brno; Petr Štourač, prof.MD.Ph.D., Study Chair — Faculty of medicince Masaryk University and University Hospital Brno
Locations (1):
- Faculty of Medicine, Masaryk University Brno, Brno, Czechia